CLINICAL TRIAL: NCT02684383
Title: A Phase 1 Evaluation of the Safety and Immunogenicity of rDEN3Δ30, a Live Attenuated Monovalent Dengue Virus Vaccine
Brief Title: Evaluation of the Safety and Immunogenicity of rDEN3Δ30, a Live Attenuated Monovalent Dengue Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 304
Record Dates: First submitted 2016-02-16; First posted 2016-02-18 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Dengue
Keywords: Dengue Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rDEN3∆30 vaccine (Experimental): Participants will receive the rDEN3∆30 vaccine at Day 0.
  Interventions: Biological: rDEN3∆30
- Placebo (Placebo Comparator): Participants will receive placebo at Day 0.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rDEN3∆30 — 10^3 plaque-forming units (PFUs); administered by subcutaneous injection in the deltoid region of the upper arm
  Arms: rDEN3∆30 vaccine
Biological: Placebo — Administered by subcutaneous injection in the deltoid region of the upper arm
  Arms: Placebo

SUMMARY:
Infection with dengue viruses is the leading cause of hospitalization and death in children in many tropical Asian countries, and the development of a dengue vaccine is a top health priority. This study will evaluate the safety and immunogenicity of a live attenuated monovalent dengue virus vaccine (rDEN3Δ30) in healthy adults with no history of previous flavivirus infection.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and immunogenicity of a live attenuated monovalent dengue virus vaccine (rDEN3Δ30) in healthy flavivirus-naive adults.

Participants will be randomly assigned to receive the rDEN3Δ30 vaccine or placebo at Day 0. Study visits will occur on Days 2, 4, 6, 8, 10, 12, 14, 16, 21, 28, 56, 90, and 180. Visits will include physical examinations and blood collection. All participants will record their temperature 3 times a day from Day 0 through Day 16. Some participants may be admitted to the clinic for an inpatient (overnight) stay during the first 16 days of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 18 and 50 years of age, inclusive.
* Good general health as determined by physical examination, laboratory screening, and review of medical history.
* Available for the duration of the study, approximately 26 weeks post-vaccination.
* Willingness and availability for potential inpatient admission in the inpatient unit following receipt of rDEN3Δ30.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Females Only: Female subjects of childbearing potential willing to use effective contraception beginning long enough before dosing to ensure method specific efficacy for the duration of the trial. Reliable methods of contraception include hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (greater than or equal to 6 months since last sexual encounter). All female subjects will be considered having childbearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria:

* Females Only: Currently pregnant, as determined by positive beta-human chorionic gonadotropin (HCG) test, or breastfeeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the requirements of the study protocol.
* Confirmed screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in this protocol. Confirmation will be obtained by repeating the test to ensure the abnormal value was not due to aberrancy.
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational or family problems, as indicated by subject history.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (emergency room visit or hospitalization within the last 6 months).
* HIV infection, by screening and confirmatory assays.
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays.
* Hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening.
* Any known immunodeficiency syndrome.
* Use of anticoagulant medications.
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination.
* Asplenia.
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination.
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis virus, or West Nile virus).
* Previous receipt of a flavivirus vaccine (licensed or experimental).
* Anticipated receipt of any investigational agent in the 28 days before or after vaccination.
* Subject has definite plans to travel to a dengue-endemic area during the study.
* Known allergy to antipyretics.
* Refusal to allow storage of specimens for future research.

Other Treatments and Ongoing Exclusion Criteria:

The following criteria will be reviewed on days 28 and 56 post-vaccination. If any become applicable during the study, then the subject will not be included in further immunogenicity evaluations, as of the exclusionary visit. The subject will, however, be encouraged to remain in the study for safety evaluations for the duration of the study.

Ongoing Exclusion Criteria:

* Use of any investigational drug or investigational vaccine other than the study vaccine during the 28-day period post-vaccination.
* Chronic administration (greater than or equal to 14 days) of steroids (defined as prednisone equivalent of greater than or equal to 10 mg per day), immunosuppressants, or other immune-modifying drugs initiated during the 28-day period post-vaccination (topical and nasal steroids are allowed).
* Receipt of a licensed vaccine during the 28-day period post vaccination.
* Receipt of immunoglobulins and/or any blood products during the 28-day period post vaccination.
* Pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related adverse events (AEs) | Measured through Day 28 post-vaccination
Level of anti-DENV-3 neutralizing antibody | Measured through Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Pierce, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Center for Immunization Research (CIR), Johns Hopkins School of Public Health, Baltimore, Maryland
  - University of Vermont Medical Center, Burlington, Vermont